CLINICAL TRIAL: NCT06809998
Title: COSTI: COntralateral CorticoSTeroid Injection in Total Knee Arthroplasty - A Triple Blinded, Randomized Controlled Trial Pilot Study
Brief Title: COntralateral CorticoSTeroid Injection in Total Knee Arthroplasty
Acronym: COSTI
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Unity Health Toronto (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: 24-158
Record Dates: First submitted 2025-01-20; First posted 2025-02-05 (Actual); Last update posted 2025-12-18 (Actual); Status verified 2025-01

CONDITIONS: Total Knee Anthroplasty; Osteoarthritis(Primary); Osteoarthritis (OA) of the Knee; Bilateral Knee Osteoarthritis
Keywords: COSTI; Total Knee Arthroplasty; Corticosteroid Injection
MeSH Terms: conditions — Osteoarthritis | interventions — Adrenal Cortex Hormones; Methylprednisolone; Bupivacaine; Epinephrine

STUDY DESIGN:
Intervention Model Description: Triple-blind randomized controlled superiority trial
Who Masked: Participant, Care Provider, Outcomes Assessor
Masking Description: This trial will be triple-blinded, meaning none of the patient, the treating most responsible surgeon or the outcome assessors (i.e. advanced practice physical therapists) will be aware of the treatment allocation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A - Corticosteroid Injection (Experimental): Corticosteroid injection - 80mg methylprednisolone (total volume 2ml) with 6 mL of 1% Bupivacaine without epinephrine (Total Volume 8 mL).
  The patient will be brought to the regional room where a fully licensed anaesthesiologist will perform standard of care anaesthesia followed by an ultrasound guided intra-articular knee injection with steroid AFTER the spinal neuraxial blockage has already been administered.
  Interventions: Drug: Corticosteroid Injection - 80mg methylprednisolone (total volume 2ml) with 6 mL of 1% Bupivacaine without epinephrine (Total Volume 8 mL).
- Group B - Band-Aid Placement (Sham Comparator): The patient will be brought to the regional room where a fellowship trained interventional pain/regional anaesthesiologist will perform standard of care anaesthesia followed by the application of a band-aid.
  Interventions: Other: Band-Aid

INTERVENTIONS:
Drug: Corticosteroid Injection - 80mg methylprednisolone (total volume 2ml) with 6 mL of 1% Bupivacaine without epinephrine (Total Volume 8 mL). — Corticosteroid Injection - 80mg methylprednisolone (total volume 2ml) with 6 mL of 1% Bupivacaine without epinephrine (Total Volume 8 mL).
  Arms: Group A - Corticosteroid Injection
Other: Band-Aid — Band-Aid
  Arms: Group B - Band-Aid Placement

SUMMARY:
Through a triple-blinded randomized control trial, the primary purpose of this pilot study is to assess the efficacy of administering peri-operative contralateral corticosteroid injection in patients undergoing TKA. The secondary outcome was to assess the effect of contralateral corticosteroid injection on pain and functional outcomes of patients undergoing TKA.

DETAILED DESCRIPTION:
Total knee arthroplasty (TKA) is a common and successful procedure used to improve the quality of life and function for patients experiencing debilitating pain from degenerative knee osteoarthritis (OA).

Some patients with knee OA have bilateral involvement and surgery may be needed in both knees. Having bilateral knee OA is a known risk factor for dissatisfaction, as there can be an overuse of the less affected, contralateral knee, in order to avoid symptoms from the more severely affected knee. Moreover, one of the principal determinants of patient-reported functional outcome after a unilateral TKA is residual pain and limited function in the contralateral, un-replaced knee.

One option to improve range of motion, pain, functional scores and reduce postoperative stiffness on both knees is a bilateral TKA; however, it has been previously reported to have a higher risk of serious cardiac complications, pulmonary complications, and mortality when compared with a unilateral TKA. A less invasive and widely available treatment option is intra-articular corticosteroids applied pre-/peri-operatively in the contralateral (un-replaced) knee to improve post-operative rehabilitation.

Intra-articular corticosteroids are extensively used to reduce inflammation and pain in inflamed arthritic joints. They are associated with a moderate improvement in pain and a small improvement in physical function usually up to 3 months after injection. The use of intra-articular corticosteroids in patients with symptomatic knee OA has been shown to improve Visual Analog Scale (VAS) scores at up to 3 months, as well as the WOMAC scores up to 6 months, compared with baseline scores. There is limited data on contralateral steroid injections and its impact on surgical site infection or PROMs.

It is estimated that from 6.5% to 20% of patients report early dissatisfaction after knee replacement surgery. Furthermore, having bilateral OA is a known risk factor for dissatisfaction among patients who undergo TKA. Residual pain, limited function and limited range of motion are primary factors in patient satisfaction after undergoing TKA. Therefore, improved pain control in the contralateral knee is hypothesized to play a role in improving patient satisfaction after a TKA on the opposite side, in addition to helping with the post-operative rehabilitation process.

Understanding whether contralateral steroid injections confer superior functional and/or patient reported outcome measures after a TKA is critical to enhance patient care and improve patient functional outcomes in OA patients. There is currently a lack of high-quality prospective trials investigating the use of contralateral corticosteroid injections for TKA outcomes.

The COSTI trial (Contralateral Steroid Injection in Total Knee Arthroplasty) was developed to fill this knowledge gap. We propose a prospective, triple-blinded (patient, surgeon and outcome assessor), randomized controlled trial comparing contralateral corticosteroid knee injections versus placing a band-aid (control) in patients with bilateral osteoarthritis undergoing a TKA for osteoarthritis.

ELIGIBILITY:
Inclusion Criteria:

* Patients 18 years of age and older
* Primary osteoarthritis diagnosis with indication for primary elective unilateral TKA
* No previous contralateral knee injections (steroids/biologics) within one year of study
* Not scheduled for bilateral TKA or a subsequent staged contralateral TKA within the next six months
* No previous or active infection or trauma (osseous/ligamentous/extensor mechanism) on the contralateral knee
* Contralateral knee pain & symptoms - defined as a VAS of >4/10 at initial pre-op visit
* Contralateral knee OA quantified as: Kellgren and Lawrence grade >2-4

  * Assessed by PI (AK) who will not be contributing any patients to the study through examination of blinded knee radiographs (3 views: AP/lateral/Sunrise)
* Patient is able to read and understand English and provide informed consent to participation in the study

Exclusion Criteria:

* Other aetiologies of OA that warrants TKA (inflammatory or post traumatic arthritis)
* Cognitive impairment (dementia, Alzheimer's, uncontrolled delirium) which will prevent patients from completing primary outcome measure or comply with follow-up requirements
* Previous TKA or ORIF or nailing on either knee
* Previous or active knee infection or extensor mechanism disruption
* Previous arthroscopy on either knee
* Medical contraindication to elective TKA surgery

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-01-24 (Actual); Primary Completion 2026-04-30 (Estimated); Study Completion 2027-04-30 (Estimated)

PRIMARY OUTCOMES:
Oxford Knee Score (OKS) | 4-, 8-, 12-weeks and 1-year post-surgery
  Repeated mean score of a short questionnaire consisting of 12 questions ranging from 0 to 48 points, designed to assess function and pain after knee replacement surgery. Higher values represent a better outcome.

SECONDARY OUTCOMES:
Visual Analogue Scale (VAS) Pain Score | 4-, 8-, 12-weeks and 1-year post-surgery
  Assess pain from a visual scale that ranges from 0 to 10. Straight line with the endpoints defining extreme limits such as 'no pain at all' (zero) and 'pain as bad as it could be' (ten). Assess both the operative and injected knees.
EuroQol five-dimensional descriptive system (EQ-5D-5L) | 4-, 8-, 12-weeks and 1-year post-surgery
  The European Quality of Life 5 Dimensions (EQ5D) is a patient reported outcome where patients self rate their level of severity of health status and health related quality of life. Consists of 5 dimensions (mobility, selfcare, usual activities, pain/discomfort, anxiety/depression) and each one of them has 5 levels (no problems, slight problems, moderate problems, severe problems, and extreme problems) where patients will indicate how they feel regarding their health status and quality of life.
Knee range of motion (ROM) | 4-, 8-, 12-weeks and 1-year post-surgery
  The therapist/assessor uses a goniometer (instrument that measures an angle of a joint) to measure the degree of knee flexion and extension of a patient. Knee ROM of both the operated and injected knees will be taken.
  Knee Flexion - the measurable degree in which the leg (and knee joint) is bent. Knee Extension - The measurable degree in which the knee is extended (making the joint angle larger, or straightening the knee.
Timed Up Go Test (TUG) | 4-, 8-, 12-weeks and 1-year post-surgery
  TUG is a simple test used to assess a person's mobility (in seconds) and requires both static and dynamic balance. A line is placed on the floor 3 meters away from a chair where patient will be sitting.
  When instructed to "GO" patient will stand, walk to a line on the floor at his/her regular pace, turn around and walk back to the chair and sit down. The longer it takes for subject to complete the test, higher is the risk of fall and lower is the its functional mobility.
  Reference values are:
  60-69 years old = 8.1 seconds; 70-79 years old = 9.2 seconds; 80-99 years old = 11.3 seconds. Over 14 seconds is associate with high risk of fall
Forgotten Joint Score (FJS) | 12-weeks and 1-year post-surgery
  A patient-reported outcome measure (PROM) that assesses how well a patient can forget about an affected knee after surgery. 12-question survey that asks patients to rate their awareness of their knee during daily activities.
  Patients answer each question on a scale of 0-4, with 0 being "never aware" and 4 being "mostly aware". The final score ranges from 0-100, with higher scores indicating less awareness of the knee.

OTHER OUTCOMES:
Feasibility - recruitment | 1.5 years
  Ability to recruit 60 patients.

CONTACTS AND LOCATIONS:
Overall Officials: Amir Khoshbin, MD, FRCS (C), Principal Investigator — Unity Health Toronto
Locations (1):
- St. Michael's Hospital, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Matzkin EG, Curry EJ, Kong Q, Rogers MJ, Henry M, Smith EL. Efficacy and Treatment Response of Intra-articular Corticosteroid Injections in Patients With Symptomatic Knee Osteoarthritis. J Am Acad Orthop Surg. 2017 Oct;25(10):703-714. doi: 10.5435/JAAOS-D-16-00541. PMID 28953085
- [Background] da Costa BR, Hari R, Juni P. Intra-articular Corticosteroids for Osteoarthritis of the Knee. JAMA. 2016 Dec 27;316(24):2671-2672. doi: 10.1001/jama.2016.17565. PMID 28027351
- [Background] Tian K, Cheng H, Zhang J, Chen K. Intra-articular injection of methylprednisolone for reducing pain in knee osteoarthritis: A systematic review and meta-analysis. Medicine (Baltimore). 2018 Apr;97(15):e0240. doi: 10.1097/MD.0000000000010240. PMID 29642145
- [Background] Fu D, Li G, Chen K, Zeng H, Zhang X, Cai Z. Comparison of clinical outcome between simultaneous-bilateral and staged-bilateral total knee arthroplasty: a systematic review of retrospective studies. J Arthroplasty. 2013 Aug;28(7):1141-7. doi: 10.1016/j.arth.2012.09.023. Epub 2013 Mar 19. PMID 23518424
- [Background] Restrepo C, Parvizi J, Dietrich T, Einhorn TA. Safety of simultaneous bilateral total knee arthroplasty. A meta-analysis. J Bone Joint Surg Am. 2007 Jun;89(6):1220-6. doi: 10.2106/JBJS.F.01353. PMID 17545424
- [Background] Sheth DS, Cafri G, Paxton EW, Namba RS. Bilateral Simultaneous vs Staged Total Knee Arthroplasty: A Comparison of Complications and Mortality. J Arthroplasty. 2016 Sep;31(9 Suppl):212-6. doi: 10.1016/j.arth.2016.03.018. Epub 2016 Mar 17. PMID 27430183
- [Background] Bagsby D, Pierson JL. Functional outcomes of simultaneous bilateral versus unilateral total knee arthroplasty. Orthopedics. 2015 Jan;38(1):e43-7. doi: 10.3928/01477447-20150105-59. PMID 25611419
- [Background] Meehan JP, Monazzam S, Miles T, Danielsen B, White RH. Postoperative Stiffness Requiring Manipulation Under Anesthesia Is Significantly Reduced After Simultaneous Versus Staged Bilateral Total Knee Arthroplasty. J Bone Joint Surg Am. 2017 Dec 20;99(24):2085-2093. doi: 10.2106/JBJS.17.00130. PMID 29257014
- [Background] Gunaratne R, Pratt DN, Banda J, Fick DP, Khan RJK, Robertson BW. Patient Dissatisfaction Following Total Knee Arthroplasty: A Systematic Review of the Literature. J Arthroplasty. 2017 Dec;32(12):3854-3860. doi: 10.1016/j.arth.2017.07.021. Epub 2017 Jul 21. PMID 28844632
- [Background] Clement ND, Bardgett M, Weir D, Holland J, Gerrand C, Deehan DJ. The rate and predictors of patient satisfaction after total knee arthroplasty are influenced by the focus of the question: a standard satisfaction question is required. Bone Joint J. 2018 Jun 1;100-B(6):740-748. doi: 10.1302/0301-620X.100B6.BJJ-2017-1292.R1. PMID 29855236
- [Background] Huang S, Li X, Tang Y, Stiphan S, Yan B, He P, Xu D. Different patient satisfaction levels between the first and second knee in the early stage after simultaneous bilateral total knee arthroplasty (TKA): a comparison between subjective and objective outcome assessments. J Orthop Surg Res. 2017 Jul 26;12(1):121. doi: 10.1186/s13018-017-0605-0. PMID 28747231
- [Background] Walmsley P, Murray A, Brenkel IJ. The practice of bilateral, simultaneous total knee replacement in Scotland over the last decade. Data from the Scottish Arthroplasty Project. Knee. 2006 Mar;13(2):102-5. doi: 10.1016/j.knee.2006.01.003. Epub 2006 Feb 14. PMID 16481171
- [Background] Marmon AR, Zeni JA Jr, Snyder-Mackler L. Perception and presentation of function in patients with unilateral versus bilateral knee osteoarthritis. Arthritis Care Res (Hoboken). 2013 Mar;65(3):406-13. doi: 10.1002/acr.21825. PMID 22933450
- [Background] Noble PC, Conditt MA, Cook KF, Mathis KB. The John Insall Award: Patient expectations affect satisfaction with total knee arthroplasty. Clin Orthop Relat Res. 2006 Nov;452:35-43. doi: 10.1097/01.blo.0000238825.63648.1e. PMID 16967035
- [Background] Lim JB, Chou AC, Chong HC, Lo NN, Chia SL, Tay KJ, Yeo SJ. Are patients more satisfied and have better functional outcome after bilateral total knee arthroplasty as compared to total hip arthroplasty and unilateral total knee arthroplasty surgery? A two-year follow-up study. Acta Orthop Belg. 2015 Dec;81(4):682-9. PMID 26790791